CLINICAL TRIAL: NCT01176552
Title: Granulocyte-macrophage Colony-stimulating Factor, Interferon Alpha and Interleukin-2 as Adjuvant Treatment for High-risk Renal Cell Carcinoma
Brief Title: Granulocyte-macrophage Colony-stimulating Factor, Interferon and Interleukin-2 as Adjuvant Treatment for Renal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kidney Cancer Research Bureau (Other)
Responsible Party: Lev Demidov, N.N. Blokhin Russian Cancer Research Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1114-6557
Record Dates: First submitted 2010-04-13; First posted 2010-08-06 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Renal Cell Carcinoma
Keywords: Kidney Cancer; Renal cell carcinoma; High risk; Adjuvant therapy
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Interferon-alpha; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study group: GM-CSF, IFN, IL-2 (Experimental)
  Interventions: Drug: GM-CSF, IFN alpha and IL-2

INTERVENTIONS:
Drug: GM-CSF, IFN alpha and IL-2 — Treatment during 6 months: GM-CSF, 1 mcg/kg, 3 times per week, subcutaneously, first week of each month; IFN, 10 MIU, 3 times per week, subcutaneously, second week, and IL-2, 1 MIU, 3 tiw, intravenously, third week. Fourth week of each month was free from treatment.

SUMMARY:
This prospective study assesses toxicity and potential efficacy of granulocyte-macrophage colony-stimulating factor (GM-CSF), interferon (IFN) alpha and interleukin-2 (IL-2) postoperatively in patients with high-risk renal cell carcinoma (RCC).

DETAILED DESCRIPTION:
Patients with high-risk RCC have a dismal prognosis. To date, no effective adjuvant therapy exists for this patients category. We suggest that combination of granulocyte-macrophage colony-stimulating factor (GM-CSF), interferon alpha (IFN) and interleukin-2 (IL-2) stimulate immune system from dendritic cells till cytotoxic T-lymphocytes step by step and eliminate residuary tumor cells.

This prospective, non-randomized, phase II trial assessed low-dose GM-CSF, IFN and IL-2 postoperatively in patients with high-risk renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* completely resected advanced high-risk RCC
* T3b-c, T4, or N1-2, or M1 disease resected to no evidence of disease (AJCC-TNM, 2002) Patients must have recovered from any effects of surgery, which must have been - excellent performance status (Eastern Cooperative Oncology Group performance status of 0 or 1);
* adequate organ function defined as WBC count 4,000/µL, platelet count 100,000/µL, hemoglobin 10 g/dL, serum creatinine 1.5 mg/dL or creatinine clearance 60 mL/min, and direct bilirubin 1.5 mg/dL; and forced expiratory volume at 1 second more than 2.0 L or 75% of predicted for height and age from pre-enrollment pulmonary function testing
* age 18 years and older

Exclusion Criteria:

* history or evidence of cardiac disease on ECG or autoimmunity
* prior systemic treatment for RCC
* history of invasive malignancy in the past 5 years or human immunodeficiency virus positivity
* positive pregnancy test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2004-05; Primary Completion 2008-09 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3.5 years

SECONDARY OUTCOMES:
Progression rate | 28 months
Overall survival (OS) | 5 years
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lev Demidov, M.D., D.Sc., Principal Investigator — N.N. Blokhin Russian Cancer Research Center
Locations (1):
- N.N. Blokhin Russian Cancer Research Center, Moscow, Russia